CLINICAL TRIAL: NCT06407531
Title: Examining the Effect of Virtual Reality Application on Patient's Anxiety and Vital Signs Before Colonoscopy: A Randomized Controlled Study
Brief Title: Before Colonoscopy Effect of Virtual Reality Application on Anxiety and Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Seda Cansu Yeniğün, Lecturer Dr., Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VRG208
Record Dates: First submitted 2024-05-03; First posted 2024-05-09 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Colonoscopy
Keywords: virtual reality glasses; surgical nursing; colonoscopy

STUDY DESIGN:
Intervention Model Description: 30 minutes before colonoscopy, the patients' systolic, diastolic blood pressure and heart rate were measured and recorded. Anxiety levels were determined with VAS. Afterwards, the patients were shown videos using virtual reality glasses. 5-10 minutes before the colonoscopy, the patients' systolic, diastolic blood pressure and heart rate were measured and recorded. Anxiety levels were determined with VAS.
Who Masked: Investigator, Outcomes Assessor
Masking Description: While the principal investigator and another co-researcher collected data, the co-researcher collected and recorded the data without having any knowledge of the results of the study.
  Data analysis will be completed by an independent researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-G (Experimental): The patient will wear virtual glasses and watch a video 30 minutes before the procedure.
  Interventions: Other: VR-G
- Control (No Intervention): No intervention will be performed on control group patients and the standard care protocol of the clinic will be applied.

INTERVENTIONS:
Other: VR-G — Patients watched videos with virtual glasses before undergoing colonoscopy
  Arms: VR-G

SUMMARY:
This study was planned to examine the effect of virtual reality application on the patient's anxiety and vital signs before colonoscopy. The hypotheses of the research are as follows:

H1: Virtual reality application before colonoscopy has an effect on patients' anxiety and vital signs.

H0: Virtual reality application before colonoscopy has no effect on patients' anxiety and vital signs.

Before colonoscopy, patients in the study group will be asked to watch videos using virtual reality glasses.

DETAILED DESCRIPTION:
After obtaining the ethics committee and institutional permission for the research, the researcher was taken to the hospital for the colonoscopy procedure.

He/she will introduce himself/herself to the patients and explain the purpose of the research. Patients who volunteered to participate in the study Informed consent will be obtained. Data regarding the socio-demographic characteristics of the patients included in the patient introduction form The patient will be interviewed face to face, and data regarding the patients' clinical characteristics will be recorded from the patient file. colonoscopy Data will begin to be collected from the first patient to undergo the procedure. Anxiety and life assessment with VAS 30 minutes before the procedure The findings will be considered. According to the randomization, the patient in the virtual reality glasses group was first asked by the researcher.

It will be explained to the patient that he will wear the glasses for 30 minutes and watch a video before the procedure. By researcher 30 When the minute is up, the patient will be informed and asked to remove the glasses. No intervention was made to the patient in the control group.

It will not be done. Anxiety and vital signs were measured with VAS 5-10 minutes before the procedure began in all patient groups.

will be looked into. After each patient use, the virtual reality glasses will be cleaned and dried with alcohol-based cleaning material.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Being literate,
* Be 18 years or older.

Exclusion Criteria:

* Performing colonoscopy at the same time as endoscopy,
* Using any analgesic or anxiolytic,
* Having a visual or hearing impairment,
* Performing an emergency colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Anxiety (Visual Analog Scale-Anxiety) | 30 minutes before colonoscopy
  Patients' anxiety will be evaluated (0-10 point). Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no anxiety and "10" means the most severe anxiety. In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Anxiety (Visual Analog Scale-Anxiety) | 5-10 minutes before colonoscopy
  Patients' anxiety will be evaluated (0-10 point). Grading is made with a 10 cm long horizontal or vertical ruler on the scale and "0" means no anxiety and "10" means the most severe anxiety. In the application, the patient was asked to mark the intensity of pain he felt on the ruler and the value was measured and recorded.
Systolic blood pressure | 30 minutes before colonoscopy
  In the measurement of vital signs of individuals, devices that measure digital blood pressure will be used by applying the necessary hygiene rules at patient transitions.
Systolic blood pressure | 5-10 minutes before colonoscopy
  In the measurement of vital signs of individuals, devices that measure digital blood pressure will be used by applying the necessary hygiene rules at patient transitions.
Diastolic blood pressure | 30 minutes before colonoscopy
  In the measurement of vital signs of individuals, devices that measure digital blood pressure will be used by applying the necessary hygiene rules at patient transitions.
Diastolic blood pressure | 5-10 minutes before colonoscopy
  In the measurement of vital signs of individuals, devices that measure digital blood pressure will be used by applying the necessary hygiene rules at patient transitions.
Heart rate | 5-10 minutes before colonoscopy
  In the measurement of vital signs of individuals, devices that measure digital pulse will be used by applying the necessary hygiene rules at patient transitions.
Heart rate | 30 minutes before colonoscopy
  In the measurement of vital signs of individuals, devices that measure digital pulse will be used by applying the necessary hygiene rules at patient transitions.

CONTACTS AND LOCATIONS:
Locations (1):
- Finike State Hospital, Antalya, Finike, Turkey (Türkiye)